CLINICAL TRIAL: NCT00145275
Title: To Assess the Efficacy of Over-the-counter Analgesics in the Prevention/Treatment of Transient Post-dose Symptoms Following Zoledronate Infusion in Post-menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446H2407
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Osteopenia
Keywords: zoledronic acid; bisphosphonate; Low bone mass
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
Zoledronic acid is a medicine being studied in people with low bone mass. Side effects such as headache, fever, muscle aches, and pains, may occur following the infusion. This study will investigate the use of over-the-counter medicines to improve these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than or equal to 45 years and less than or equal to 75 years of age inclusive
* Low bone mineral density

Exclusion Criteria:

* Certain prior treatments for low bone mass/osteopenia
* Current use of medicines (prescription or non-prescription) for pain, fever, or inflammation
* Impaired kidney function

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 45 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 455
Dates: Start 2004-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Temperature increase

SECONDARY OUTCOMES:
Questionnaires
VAS (visual analog scale)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Unavailable, Georgia
  - Unavailable, Illinois
  - Unavailable, Indiana
  - Unavailable, Iowa
  - Unavailable, Kansas
  - Unavailable, Washington
- Multiple, Australia
- Multiple, Canada
- Multiple, Russia
- Multiple, South Africa